CLINICAL TRIAL: NCT06526065
Title: Molecular Mechanisms in Malignant Lymphoma- Predict
Brief Title: Molecular Mechanisms in Malignant Lymphoma- Predict (MMML Predict)
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Collaborators: Charite University, Berlin, Germany (Other); Wuerzburg University Hospital (Other); University Hospital Ulm (Other); University of Leipzig (Other); University Hospital Regensburg (Other); University Hospital Freiburg (Other); Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); University of Kiel (Other); University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Trümper, Prof. Dr. Lorenz Trümper, University Medical Center Goettingen
Other Study IDs: 4/3/24
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Leucocytes Liquid Biopsy Tumor paraffin embedded biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The trial aims at the construction and validation of an accurate, affordable and simple prognostic tool to be used in everyday clinical practice, which allows the early and reliable identification of DLBCL patients who have a very high risk of treatment failure following R-CHOP/-like first-line therapy.

DETAILED DESCRIPTION:
Observational study of 500 recruited and 300 evaluable patients with de novo large cell B Cell lymphoma, age 18-80. Standard guideline recommended treatment by treating physicians discretion. Collection of clinical data, PET-CT data, liquid biopsy, WGSequencing to determine optimal prognostic factors to surpass prediction offered by current IPI.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of DLBCL&LBCL
2. Planned treatment with guideline-based first-line therapy
3. Patient's consent
4. All genders, Patient age ≥ 18 years
5. Ability to consent

Exclusion Criteria:

1. Treatment with R-CHOP/-like regimens already started
2. Relationship of dependence/ direct employment with the investigator
3. Active HIV-infection
4. Presence history of other active cancers (with the exception of basal cell carcinoma of the skin)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with initial diagnosis of DLBCL qualified for a treatment with R-CHOP/ R-CHOP-like regime
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS-2) with 95% confidence intervals | 2 years
  PFS is defined as the time from the day of inclusion into the observation trial through one of the following events, whichever comes first:
  * Change of treatment due to response in iPET (PD - Progressive Disease)
  * Disease progression
  * Relapse
  * Death due to any cause Patients without event at the time of analysis will be censored at the most recent date of disease assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Overall Survival (OS) is defined as the time from the day of inclusion into the observation trial to death due to any cause; patients without event will be censored at the last date known to be alive.
Event-free survival (EFS) | 5 years
  Event-free survival (EFS) is defined as the time from the day of inclusion into the observation trial through one of the following events, whichever comes first:
  * Change of treatment due to response in iPET (PD)
  * Disease progression
  * Start of additional, unplanned anti-lymphoma therapy (consolidation radiotherapy as per S3LL excluded)
  * Relapse
  * Death due to any cause
Response rates | 2 years
  overall response to treatment
Safety and toxicity | 5 years
  treatment side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Trümper, Principal Investigator — PI of the study
Locations (1):
- Universitätsmedizin Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No